CLINICAL TRIAL: NCT01248429
Title: National Study of Prevalence of Creatinine Phosphokinase (CPK) Increase in Patients With Solid Tumors Treated by Inhibitors of Tyrosine Kinases (TKI)
Brief Title: Prevalence of Creatinine Phosphokinase Increase in Patients With Solid Tumors Treated by Inhibitors of Tyrosine Kinases
Acronym: TKI-CPK-1003
Status: Completed | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Other Study IDs: TKI-CPK 1003
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Cancer; Solid Tumor
Keywords: thyrosine kinase inhibitor; phosphokinase creatinin; myalgia
MeSH Terms: conditions — Neoplasms; Myalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient treated by TKI: Any patient with solid tumor and treated by Thyrosine Kinase Inhibitor for at least 1 week
  Interventions: Biological: CPK dosage; Other: Clinical exam

INTERVENTIONS:
Biological: CPK dosage — CPK dosage during a blood sample realized at least one week after the begining of the treatment
Other: Clinical exam — Examination of the patient for myalgia, cramps, medical history and concomitant medication

SUMMARY:
This study describes the elevation of CPK in patient treated for solid tumors by TKI

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid tumor treated by inhibitor of tyrosin kinase for at least 1 week
* Patient examined AND with a routine blood test planned
* Patient informed of procedure for the study who was not opposed to it

Exclusion Criteria:

* Patient treated for malignant hemopathy
* Patient no treated by inhibitor of thyrosine kinase or for less than 1 week
* Patients with no routine blood laboratory tests planned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for a solid tumor by thyrosin kinase inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the prevalence of the CPK increase | Within 3 days after a clinical exam
  Dosage of CPK during standard blood sampling. The increase of CPK is defined when CPK value > USL

SECONDARY OUTCOMES:
Correlation myalgia/CPK increase | During the clinical exam
  To determine the correlation between myalgia and CPK blood, taking into account the risk factors leading to CPK increase

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ADENIS, MD, PhD, Principal Investigator — Centre Oscar Lambret
Locations (27):
- France (27):
  - Centre Paul Papin, Angers
  - Hôpital Jean Minjoz, Besançon
  - CHU Bordeaux, Bordeaux
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Hôpital Henri Mondor - APHP, Créteil
  - Centre Oscar Lambret, Lille
  - CHU Limoges, Limoges
  - Hôpital Edouard Herriot, Lyon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hôpital Saint-Louis - APHP, Paris
  - Hôpital Cochin - APHP, Paris
  - Hôpital Tenon - APHP, Paris
  - Institut Curie, Paris
  - Institut Jean Godinot, Reims
  - CHU Robert Debré, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre René Huguenin, Saint-Cloud
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Institut Claudius Régaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif